CLINICAL TRIAL: NCT01473368
Title: Open Label, Randomized Pilot Study to Examine The Effects of the Probiotic Saccharomyces Boulardii, the Antibiotic Amoxicillin/Clavulanate and the Combination on the Gut Microbiota of Healthy Volunteers
Brief Title: Effects of S. Boulardii and Amoxicillin/Clavulanate on Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Biocodex (Industry)
Responsible Party: Principal Investigator, Ciaran Kelly, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011P000389
Record Dates: First submitted 2011-11-15; First posted 2011-11-17 (Estimated); Results first posted 2016-09-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: human Gut Microbiota; gut microbiota; gut microbiome; probiotic; antibiotic; antibiotic-associated diarrhea; intestinal bacterial overgrowth
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- prebiotic (Saccharomyces boulardii) (Active Comparator): 500 mg, 2 times daily for 14 days
  Interventions: Dietary Supplement: Saccharomyces boulardii
- antibiotic (Amoxicillin Clavulanate) (Active Comparator): 875/125 mg 2 times daily at least 1 hour before meals for 7 days
  Interventions: Drug: Amoxicillin Clavulanate
- combination (prebiotic and antibiotic) (Active Comparator): Amoxicillin Clavulanate for 7 days (days 1 to 7; 875/125 mg 2 times daily at least 1 hour before meals) in addition to the dietary supplement Saccharomyces boulardii for 14 days (days 1 to 14; 500 mg, 2 times daily).
  Interventions: Dietary Supplement: Saccharomyces boulardii; Drug: Amoxicillin Clavulanate
- control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Saccharomyces boulardii — 500 mg, 2 times daily for 14 days
  Arms: combination (prebiotic and antibiotic); prebiotic (Saccharomyces boulardii)
Drug: Amoxicillin Clavulanate — 875/125 mg 2 times daily at least 1 hour before meals for 7 days
  Arms: antibiotic (Amoxicillin Clavulanate); combination (prebiotic and antibiotic)

SUMMARY:
The purpose of this study is to compare and contrast the effects of the probiotic Saccharomyces boulardii, the antibiotic amoxicillin/clavulanate and the combination on the gut microbiota of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years (male or female)
* Good general health
* Able to comply with study requirements and to provide informed consent
* For women of childbearing potential oA negative urine pregnancy test immediately prior to starting the study treatment oAgreement to comply with approved methods of contraception during the period of active study treatment (not required during follow-up)

Exclusion Criteria:

* History of organ transplantation
* Known chronic or recurrent systemic disorder associated with immunocompromise
* A history of allergy or hypersensitivity to Saccharomyces boulardii, brewer's or baker's yeast, amoxicillin, penicillins, or cephalosporins
* History of severe allergic reaction (requiring hospital admission and/or the administration of parenteral medication or associated with dyspnoea, wheezing, hypotension, loss of consciousness).
* Oral or systemic antibacterial therapy during the 3 months prior to study enrollment
* New prescription medications during the 4 weeks prior to study enrollment
* Prescription, OTC medications or supplements that are known to alter gut function or microflora (i.e. acid antisecretory drugs, probiotics) during the 4 weeks prior to study enrollment
* Active gastrointestinal disease
* Patients with a central venous catheter
* Patients taking antifungals or laxatives within 14 days of enrolment
* Patients enrolled in other clinical trials within the past 60 days
* Prior gastrointestinal surgery (apart from appendectomy or cholecystectomy)
* History of chronic constipation with passage of fewer than 3 bowel movements per week on average
* Any condition or personal circumstance that, in the opinion of the investigator, renders the subject unlikely or unable to comply with the full study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran P Kelly, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kelly CP, Chong Nguyen C, Palmieri LJ, Pallav K, Dowd SE, Humbert L, Seksik P, Bado A, Coffin B, Rainteau D, Kabbani T, Duboc H. Saccharomyces boulardii CNCM I-745 Modulates the Fecal Bile Acids Metabolism During Antimicrobial Therapy in Healthy Volunteers. Front Microbiol. 2019 Mar 4;10:336. doi: 10.3389/fmicb.2019.00336. eCollection 2019. PMID 30881353

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination (Prebiotic and Antibiotic): Saccharomyces boulardii AND Amoxicillin Clavulanate: Amoxicillin Clavulanate for 7 days (days 1 to 7; 875/125 mg 2 times daily at least 1 hour before meals) in addition to the dietary supplement Saccharomyces boulardii for 14 days (days 1 to 14; 500 mg, 2 times daily).
- Control: Control group
Period: Overall Study
Arm/Group | Prebiotic (Saccharomyces Boulardii) | Antibiotic (Amoxicillin Clavulanate) | Combination (Prebiotic and Antibiotic) | Control
Started | 14 | 12 | 15 | 12
Completed | 13 | 12 | 12 | 12
Not Completed | 1 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prebiotic (Saccharomyces Boulardii) | Antibiotic (Amoxicillin Clavulanate) | Combination (Prebiotic and Antibiotic) | Control | Total
Number analyzed (Participants) | 13 | 12 | 12 | 12 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 12 | 12 | 49
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (9.9) | 27.4 (6.6) | 34.2 (11.4) | 27.2 (4.3) | 30.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 7 | 5 | 29
  Male | 3 | 5 | 5 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 12 | 12 | 49

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal Symptom Rating Scale
Description: Mean Gastrointestinal Symptom Rating Scale scores Range from 15 to 90 Increasing score means increasing symptoms
Time Frame: Day 0
Population: Control participants were not assessed at this time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prebiotic (Saccharomyces Boulardii) | Antibiotic (Amoxicillin Clavulanate) | Combination (Prebiotic and Antibiotic)
Number analyzed (Participants) | 13 | 12 | 12
units on a scale | 18.7 (5.4) | 18.7 (3.8) | 17.3 (2.4)

2. Primary Outcome: Gastrointestinal Symptom Rating Scale
Description: Mean Gastrointestinal Symptom Rating Scale scores Range from 15 to 90 Increasing score means increasing symptoms
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prebiotic (Saccharomyces Boulardii) | Antibiotic (Amoxicillin Clavulanate) | Combination (Prebiotic and Antibiotic) | Control
Number analyzed (Participants) | 13 | 12 | 12 | 12
Units on a scale | 23.2 (8.8) | 26.9 (14.2) | 18.1 (3.0) | 19.3 (8.1)
Statistical Analysis 1: Comparison: Antibiotic (Amoxicillin Clavulanate) vs Combination (Prebiotic and Antibiotic); Test type: Superiority or Other; p = 0.026, ANOVA

3. Primary Outcome: Gastrointestinal Symptoms Response Score
Description: Mean Gastrointestinal Symptom Rating Scale scores Range from 15 to 90 Increasing score means increasing symptoms
Time Frame: Day 14
Population: Participants analyzed were those with complete data at Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prebiotic (Saccharomyces Boulardii) | Antibiotic (Amoxicillin Clavulanate) | Combination (Prebiotic and Antibiotic) | Control
Number analyzed (Participants) | 12 | 11 | 12 | 12
units on a scale | 19.3 (5.1) | 20.3 (5.9) | 16.8 (1.6) | 18.1 (4.3)

4. Primary Outcome: Gastrointestinal Symptoms Response Scale
Description: Mean Gastrointestinal Symptom Rating Scale scores Range from 15 to 90 Increasing score means increasing symptoms
Time Frame: Day 21
Population: Participants analyzed were those with complete data at Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prebiotic (Saccharomyces Boulardii) | Antibiotic (Amoxicillin Clavulanate) | Combination (Prebiotic and Antibiotic) | Control
Number analyzed (Participants) | 12 | 11 | 12 | 12
units on a scale | 19.3 (5.7) | 18.4 (5.8) | 16.5 (2.9) | 15.8 (2.3)

5. Primary Outcome: Prevalence of Escherichia in Stool
Description: Control arm was not assessed as there was no intervention for this group.
  Before Treatment: Average of Day -7 and Day 0 During Treatment: Average of Day 3, Day 7, Day 10, Day 13 After Treatment: Average of Day 21
Time Frame: Day -7 to Day 21
Measure: Mean (Standard Deviation); unit: percentage of total bacteria
Groups:
- Prebiotic (Saccharomyces Boulardii) Before Treatment: Before treatment
  Saccharomyces boulardii: 500 mg, 2 times daily for 14 days
- Prebiotic (Saccharomyces Boulardii) During Treatment: During treatment
  Saccharomyces boulardii: 500 mg, 2 times daily for 14 days
- Prebiotic (Saccharomyces Boulardii) After Treatment: After treatment
  Saccharomyces boulardii: 500 mg, 2 times daily for 14 days
Arm/Group | Prebiotic (Saccharomyces Boulardii) Before Treatment | Prebiotic (Saccharomyces Boulardii) During Treatment | Prebiotic (Saccharomyces Boulardii) After Treatment
Number analyzed (Participants) | 13 | 13 | 12
percentage of total bacteria | 0.0 (0) | 0.0 (0) | 0.1 (0)

6. Primary Outcome: Prevalence of Escherichia in Stool
Description: as for outcome 5
Time Frame: Day -7 to Day 21
Measure: Mean (Standard Deviation); unit: percentage of total bacteria
Groups:
- Antibiotic (Amoxicillin Clavulanate) Before Treatment: Before treatment
  Amoxicillin Clavulanate: 875/125 mg 2 times daily at least 1 hour before meals for 7 days
- Antibiotic (Amoxicillin Clavulanate) During Treatment: During treatment
  Amoxicillin Clavulanate: 875/125 mg 2 times daily at least 1 hour before meals for 7 days
- Antibiotic (Amoxicillin Clavulanate) After Treatment: After treatment
  Amoxicillin Clavulanate: 875/125 mg 2 times daily at least 1 hour before meals for 7 days
Arm/Group | Antibiotic (Amoxicillin Clavulanate) Before Treatment | Antibiotic (Amoxicillin Clavulanate) During Treatment | Antibiotic (Amoxicillin Clavulanate) After Treatment
Number analyzed (Participants) | 12 | 12 | 11
percentage of total bacteria | 0.1 (0) | 4.5 (0) | 0.2 (0)
Statistical Analysis 1: Comparison: Antibiotic (Amoxicillin Clavulanate) Before Treatment vs Antibiotic (Amoxicillin Clavulanate) During Treatment vs Antibiotic (Amoxicillin Clavulanate) After Treatment; Test type: Superiority or Other; p < 0.05, ANOVA

7. Primary Outcome: Prevalence of Escherichia in Stool
Description: as for outcome 5
Time Frame: Day -7 to Day 21
Measure: Mean (Standard Deviation); unit: percentage of total bacteria
Groups:
- Combination (Prebiotic and Antibiotic) Before Treatment: Before treatment
  Saccharomyces boulardii AND Amoxicillin Clavulanate: Amoxicillin Clavulanate for 7 days (days 1 to 7; 875/125 mg 2 times daily at least 1 hour before meals) in addition to the dietary supplement Saccharomyces boulardii for 14 days (days 1 to 14; 500 mg, 2 times daily).
- Combination (Prebiotic and Antibiotic) During Treatment: During treatment
  Saccharomyces boulardii AND Amoxicillin Clavulanate: Amoxicillin Clavulanate for 7 days (days 1 to 7; 875/125 mg 2 times daily at least 1 hour before meals) in addition to the dietary supplement Saccharomyces boulardii for 14 days (days 1 to 14; 500 mg, 2 times daily).
- Combination (Prebiotic and Antibiotic) After Treatment: After treatment
  Saccharomyces boulardii AND Amoxicillin Clavulanate: Amoxicillin Clavulanate for 7 days (days 1 to 7; 875/125 mg 2 times daily at least 1 hour before meals) in addition to the dietary supplement Saccharomyces boulardii for 14 days (days 1 to 14; 500 mg, 2 times daily).
Arm/Group | Combination (Prebiotic and Antibiotic) Before Treatment | Combination (Prebiotic and Antibiotic) During Treatment | Combination (Prebiotic and Antibiotic) After Treatment
Number analyzed (Participants) | 12 | 12 | 12
percentage of total bacteria | 0.0 (0) | 2.9 (0) | 0.2 (0)

8. Primary Outcome: Operational Taxonomic Units
Description: Core Microbiome includes control samples and baseline samples (Day -7 and Day 0) for antibiotic, probiotic, and combination groups. Data for Core microbiome for individual arms are not available.
  Before Treatment: Average of Day -7 and Day 0 During Treatment: Average of Day 3, Day 7, Day 10, Day 13 After Treatment: Average of Day 21
Time Frame: Day 0 to Day 21
Measure: Mean (Standard Deviation); unit: units
Groups:
- Core Microbiome: Core Microbiome
Arm/Group | Combination (Prebiotic and Antibiotic) During Treatment | Combination (Prebiotic and Antibiotic) After Treatment | Antibiotic (Amoxicillin Clavulanate) During Treatment | Antibiotic (Amoxicillin Clavulanate) After Treatment | Core Microbiome | Prebiotic (Saccharomyces Boulardii) During Treatment | Prebiotic (Saccharomyces Boulardii) After Treatment
Number analyzed (Participants) | 13 | 12 | 12 | 11 | 49 | 12 | 12
units | 449.8 (210.1) | 509.9 (251.9) | 461.1 (228.2) | 668.8 (188.4) | 730.9 (240.4) | 776.7 (167.6) | 776.7 (749.1)

ADVERSE EVENTS:
Arm/Group | Prebiotic (Saccharomyces Boulardii) | Antibiotic (Amoxicillin Clavulanate) | Combination (Prebiotic and Antibiotic) | Control
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/13 | 6/12 | 2/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prebiotic (Saccharomyces Boulardii) (N=13) | Antibiotic (Amoxicillin Clavulanate) (N=12) | Combination (Prebiotic and Antibiotic) (N=12) | Control (N=12)
Abdominal distension (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1
diarrhea (Gastrointestinal disorders) | 1 | 3 | 1 | 0
dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 1
gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 2 | 0 | 0
infrequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0
regurgitation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
vulvovaginal rash (Reproductive system and breast disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes